CLINICAL TRIAL: NCT01027195
Title: Evaluation of the Efficacy of the Bipolar Sealer Aquamantys 6.0 in Patients Undergoing Total Hip Arthroplasty
Acronym: Hip
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Salient Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-615; NCT01448967 (obsolete NCT alias)
Record Dates: First submitted 2009-12-03; First posted 2009-12-07 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-10

CONDITIONS: Hip Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Bovie Electrocautery (Placebo Comparator): Standard Bovie electrocautery [Valleylab, Boulder, Colorado] used on surgical site during primary total hip arthroplasty to deliver high frequency electrical current to seal tissues and blood vessels.
  Interventions: Device: Standard Bovie Electrocautery
- Bipolar Radiofrequency (Experimental): Aquamantys 6.0 bipolar sealer [Salient Surgical Technologies, Portsmouth, New Hampshire] used on surgical site during primary total hip arthroplasty to deliver radiofrequency energy coupled with saline solution irrigation for hemostatic sealing (i.e. shrinking of collagen in the walls of tissue vessels) at lower temperatures (<100 degrees Celsius) than standard Bovie electrocautery.
  Interventions: Device: Bipolar Radiofrequency (Aquamantys 6.0)

INTERVENTIONS:
Device: Bipolar Radiofrequency (Aquamantys 6.0)
  Other Names: Aquamantys 6.0
  Arms: Bipolar Radiofrequency
Device: Standard Bovie Electrocautery
  Arms: Standard Bovie Electrocautery

SUMMARY:
The present prospective, single-center, clinical trial is designed to evaluate the hemostatic efficacy of the hemostatic sealer Aquamantys 6.0™ in patients managed with total hip arthroplasty (THA). It is hypothesized that Aquamantys 6.0™ can improve hemostasis following total hip arthroplasty. Comparison of the functional and clinical results between THA patients having been exposed to Aquamantys 6.0™ versus a control group will be analyzed using several outcome measures including the Harris Hip Score and a pain scale. The primary variable of interest is transfusion requirements - specifically, number of patients managed with blood transfusion during the hospital stay after surgery. However, of secondary interest will be: 1) number of units transfused, 2) estimated intraoperative total blood loss, 3) change in pre- and post-operative hemoglobin levels, 4) total narcotic usage during hospital stay, 5) length of stay, 6) functional and pain outcomes (Harris Hip Score and Pain Scale), and 7) adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 85 years
* Sex: Both male and female will be included. The male-to-female ratio will depend upon the patient population.
* Stable Health: At the time of surgery based on physical examination and medical history.
* Patient exhibited preoperative radiographic evidence of joint degeneration consistent with THA that could not have been treated in non-operative fashion.
* Patient had severe hip pain and disability due to degenerative joint disease.
* Patient or patient's legal representative has signed the Informed Consent form. The patient is capable of making informed decisions regarding his/her healthcare.

Exclusion Criteria:

* Patients with history of cardiac disease, liver disease or renal disease. Severe cardiac disease, liver disease and renal dysfunction can confound different parameters within this study. Patients with decreased cardiac function from prior myocardial infarction, cardiomyopathy or congestive heart failure will likely require transfusions with packed red blood cells at lower thresholds relative to healthy counterparts for cardioprotection. Therefore, patients with a prior history of myocardial infarction, cardiomyopathy, congestive heart failure or other significant cardiac history will be excluded from this study. In addition, patients with liver dysfunction from cirrhosis or hepatitis may have impaired production of factors in the clotting cascade which may make these individuals more prone to bleed, especially with the use of anticoagulants such as lovenox. For this reason, these patients will also be excluded from this study. Finally, individuals with renal dysfunction will have decreased creatinine clearance, which may artificially elevate the levels of lovenox, thereby promoting bleeding. In addition, individuals with severe renal disease may also have associated anemia which would complicate the transfusion threshold. For this reason, individuals with chronic renal failure, diabetic nephropathy, or decreased creatinine clearance will be excluded from this study.
* Patients predonating autologous blood.
* Patients with preoperative hemoglobin level less than 11.5 g/dL or a hematocrit less than 35%. Patients with a preoperative platelet count of less than 100,000.
* Patients undergoing bilateral or revision surgery.
* Evidence of bleeding or metabolic - based hemolytic disorder (hemophilia or anticoagulation use)
* Previous history of infection in the affected joint.
* Peripheral vascular disease.
* Patient was a poor compliance risk - treated for ethanol or drug abuse, physical or mental handicap, etc.
* Patients whose personal beliefs exclude the use of blood transfusions (example: Jehovah's witness).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-08; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wael K Barsoum, MD, Principal Investigator — The Cleveland Clinic

REFERENCES:
- [Result] Barsoum WK, Klika AK, Murray TG, Higuera C, Lee HH, Krebs VE. Prospective randomized evaluation of the need for blood transfusion during primary total hip arthroplasty with use of a bipolar sealer. J Bone Joint Surg Am. 2011 Mar 16;93(6):513-8. doi: 10.2106/JBJS.J.00036. PMID 21411700

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Started | 71 | 69
Completed | 71 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery | Total
Number analyzed (Participants) | 71 | 69 | 140
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.9) | 55.7 (11.0) | 55.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 31 | 66
  Male | 36 | 38 | 74
Body-Mass Index [Mean (Standard Deviation); unit: kg/m2]
  Females | 28.6 (7.1) | 29.2 (6.1) | 28.9 (6.6)
  Males | 29.4 (4.7) | 30.4 (5.1) | 29.9 (4.9)
Baseline Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 14.6 (1.3) | 14.2 (1.2) | 14.4 (1.3)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Units Transfused
Time Frame: daily during hospital stay (an expected average of 4 days)
Measure: Mean (Standard Deviation); unit: units of blood
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Number analyzed (Participants) | 71 | 69
units of blood | 0.38 (0.83) | 0.44 (0.98)

2. Primary Outcome: Number of Patients Managed With Blood Transfusion
Time Frame: daily during hospital stay (an expected average of 4 days)
Measure: Number; unit: participants
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Number analyzed (Participants) | 71 | 69
participants | 15 | 14

3. Secondary Outcome: Estimated Blood Loss
Time Frame: Intraoperative (day of surgery)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Number analyzed (Participants) | 71 | 69
mL | 315.2 (203.4) | 368.5 (277.8)

4. Secondary Outcome: Change in Hemoglobin Level
Description: Change in hemoglobin level from baseline to the day of hospital discharge.
Time Frame: within 30 days before surgery (preop), day of hospital discharge
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Number analyzed (Participants) | 71 | 69
g/dL | -5.4 (1.6) | -5.3 (1.8)

5. Secondary Outcome: Total Narcotic Usage (Morphine-equivalent mg) During Hospital Stay
Description: Sum of daily morphine-equivalent mg narcotic usage during hospital stay.
Time Frame: daily during hospital stay (an expected average of 4 days)
Measure: Mean (Standard Deviation); unit: total morphine-equivalent mg
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Number analyzed (Participants) | 71 | 69
total morphine-equivalent mg | 156.1 (130.2) | 164.9 (123.4)

6. Secondary Outcome: Length of Stay
Time Frame: day of hospital discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Number analyzed (Participants) | 71 | 69
days | 3.3 (1.1) | 3.4 (1.6)

7. Secondary Outcome: Harris Hip Score (Outcome Score)
Description: A scoring system used to evaluate the outcome after total hip replacement. Domains include pain (44 points), function (47 points), deformity (4 points), and range of motion (5 points). A total score is computed by summing the individual domain scores, with a maximum of 100 points. Higher values represent better outcomes. A total Harris Hip Score below 70 points is generally considered a poor result, 70 to 80 fair, 80 to 90 good, and 90 to 100 excellent.
Time Frame: within 30 days before surgery (preop), 4 weeks after surgery, 12 weeks after surgery
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Number analyzed (Participants) | 71 | 69
points on a scale
  Preoperative | 59.0 (12.2) | 60.4 (11.6)
  4 Weeks Postoperative | 78.4 (9.8) | 78.4 (11.2)
  12 Weeks Postoperative | 92.8 (8.2) | 95.1 (5.4)

8. Secondary Outcome: Pain Score Scale
Description: A single scoring system used to evaluate overall pain on a scale of integers 0 to 10, with 0 representing "no pain" and 10 representing "unbearable pain." Thus, in this context, lower values represent better outcomes.
Time Frame: within 30 days before surgery (preop), 4 weeks after surgery, 12 weeks after surgery
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Number analyzed (Participants) | 71 | 69
points on a scale
  Preoperative | 6.2 (2.2) | 6.4 (2.0)
  4 Weeks Postoperative | 1.7 (1.7) | 1.7 (1.8)
  12 Weeks Postoperative | 1.2 (1.7) | 0.9 (1.2)

ADVERSE EVENTS:
Arm/Group | Bipolar Radiofrequency | Standard Bovie Electrocautery
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/69
Other Adverse Events (participants affected / at risk) | 2/71 | 4/69
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bipolar Radiofrequency (N=71) | Standard Bovie Electrocautery (N=69)
Deep Infection (Infections and infestations) | 0 (0) | 1 (1)
Coronary Ischemic Event (Cardiac disorders) | 1 (1) | 1 (1)
Deep-Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes